CLINICAL TRIAL: NCT06301230
Title: The PLET Study: A Randomized Controlled Trial of Home- Versus Hospital-based Surgical Training
Brief Title: Home- vs. Hospital-based Surgical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarunis - Universitäres Bauchzentrum Basel (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLET-2022
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Surgical Training
Keywords: Surgical training; Surgical skill performance; PLET; Portable Laparoscopic Trainer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-based surgical training group (Active Comparator): This group represents the surgical residents who trained with PLET at the hospital.
  Interventions: Device: Portable Laparoscopic Trainer (PLET)
- Home-based surgical training group (Experimental): This group represents the surgical residents who trained with PLET at home.
  Interventions: Device: Portable Laparoscopic Trainer (PLET)

INTERVENTIONS:
Device: Portable Laparoscopic Trainer (PLET) — The PLET trainer is light and easy to transport packed in a bag and consists of a foldable plastic box, which can be assembled in less than 30 seconds by means of simple handles. There are three accesses for the surgical instruments (ports) as well as a central recess over which a tablet with an integrated camera can be placed.
  Each participant received a previously prepared opaque envelope containing a black or white USB stick from the Principal Investigator with the assignments on it as part of the randomization process. The outcome assessors were blinded to the allocation.

SUMMARY:
The purpose of this study was to assess the effect of training with a personal, portable laparoscopic endo-trainer (PLET) on residents' laparoscopic skills. All participants were randomised to either a home- or hospital-based PLET training group and surgical skill performance was assessed using five laparoscopic exercises. Endpoints consisted ofsubjective and objective assessment ratings as well as exercise time and qualitative data up to 12 weeks. The primary outcome was the difference in exercise time and secondary outcomes included performance scores as well as qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* surgical resident

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Exercise time | Baseline, 6 weeks, 12 weeks
  Amount of time surgical residents need for laparoscopic exercises
Assessment rating | Baseline, 6 weeks, 12 weeks
  Subjective and objective assessment ratings of surgical skills during exercise

SECONDARY OUTCOMES:
Qualitative feedback | 12 weeks
  Open questions about motivation of participating in the study and improving surgical skills

CONTACTS AND LOCATIONS:
Locations (1):
- Clarunis Universitäres Bauchzentrum Basel, Basel, Switzerland

REFERENCES:
- [Derived] Kuemmerli C, Linke K, Daume D, Germann N, Peterli R, Muller-Stich B, Klasen JM. The PLET (Portable Laparoscopic Endo-Trainer) study: a randomized controlled trial of home- versus hospital-based surgical training. Langenbecks Arch Surg. 2024 Jun 13;409(1):186. doi: 10.1007/s00423-024-03375-z. PMID 38869683